CLINICAL TRIAL: NCT07278427
Title: Reducing Parental Substance Use, Improving Child Health Outcomes, and Enhancing Family Resilience Among Rural Families Through Ohio START (Sobriety, Treatment, and Reducing Trauma)
Brief Title: Reducing Parental Substance Use and Enhancing Family Resilience Among Rural Families Through Ohio START
Acronym: Ohio START
Status: Not yet recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Susan Yoon, Associate Professor, Ohio State University
Other Study IDs: 1R01HD119145 (NIH); 1R01HD119145-01 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorder (SUD); Rural Health; Family Resilience; Child Maltreatment; Child Well-beiing; Substance Use Recovery
Keywords: Substance use disorder; Child abuse and neglect; Rural health; Child welfare services; Low socioeconomic status; Rurality; Longitudinal study; Prospective study; Family resilience; Social network; Activity spaces; Child maltreatment; Parental substance use; Family peer mentors; Social networks; Rural families; Ohio START; Child well-being; Substance use treatment services; Family health; The START model
MeSH Terms: conditions — Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rural parents receiving Ohio START services: Parents who have entered the child welfare system due to co-occurring parental substance use and child maltreatment and who are currently enrolled in Ohio START (Ohio Sobriety, Treatment, and Reducing Trauma). The study is conducted in the context of Ohio START, a children-services-led initiative and evidence-informed intervention model currently operating in 57 counties in the state of Ohio. If both parents from the same family receive the Ohio START intervention, both are eligible to participate.
  Interventions: Behavioral: Ohio START (Ohio Sobriety, Treatment, and Reducing Trauma)

INTERVENTIONS:
Behavioral: Ohio START (Ohio Sobriety, Treatment, and Reducing Trauma) — Ohio START launched in 2017 in response to the opioid epidemic and is led by the Public Children Services Association of Ohio (PASCO). Ohio START integrates child welfare and substance use treatment systems to enhance access to treatment for parents who come into the child welfare system with addictions. Ohio START capitalizes on collaboration between the child welfare system and behavioral health providers in order to reduce parent wait times for treatment for referrals, increase parent engagement and retention in treatment, and enhance coordination of resources and support for parents and children. Another key aspect of START is the use of family peer mentors as a social network intervention. Parents are paired with family peer mentors who, through weekly visits, support participating families and enhance coordination of resources. Family peer mentors are required to have a minimum of a weekly face-to-face visit with parents for 90 days.

SUMMARY:
The goal of this observational study is to learn about the roles played by parental activity spaces and social networks in reducing parental substance use and promoting child and family health outcomes in the context of Ohio START (Sobriety, Treatment, and Reducing Trauma) for families in rural areas. This study will investigate if substance use treatment service referrals and family peer mentoring services provided by Ohio START lead to positive changes in parental activity spaces and social networks, and if these positive changes lead to better child and family outcomes. The main questions it aims to answer are:

* Does having behavioral health services (referred by Ohio START workers) close to where parents spend their time help with substance use recovery and child health?
* Does peer mentor support through Ohio START help parents build stronger social connections and family resilience, and does this lead to better long-term family health?
* Do these associations differ in rural areas compared to urban areas?

Participants will:

* Answer survey questions about their substance use, parenting, child health, and family well-being across three waves (Wave 1: when they enroll in the study, Wave 2: 6-month follow-up, and Wave 3: 12-month follow-up)
* Share information about places they go regularly (such as work, stores, and healthcare visits)
* Share information about people in their support network

DETAILED DESCRIPTION:
Co-occurring parental substance use disorder (SUD) and child maltreatment are key risk factors associated with poor health outcomes among children and families in rural areas. Importantly, rural communities face geographic, economic, and social challenges that limit their access to SUD treatment services. Ohio Sobriety, Treatment, and Reducing Trauma (Ohio START) is a family-centered child welfare service delivery intervention that builds on cross-system collaboration with behavioral health service organizations to provide timely access to SUD treatment services for parents involved with the child welfare system. Ohio START also supports parents' journey to SUD recovery through family peer mentors -individuals with lived experience in SUD recovery and previous child welfare involvement- who offer intensive recovery support. When Ohio START child welfare caseworkers refer parents to SUD treatment services located within or near the places parents regularly visit (i.e., activity spaces), parents may be more likely to engage in treatment consistently and experience improvements in their health and family well-being. Similarly, when parents actively engage with family peer mentors, who help them connect with treatment and recovery communities, they may experience positive shifts in their activity spaces and social networks. Yet, it remains unclear how access to SUD treatment services within parents' activity spaces and greater engagement with family peer mentors influence child and family health outcomes, especially among low-income families in rural areas. These are important questions that, if answered, could enhance interventions to better serve families in rural communities. Capitalizing on a unique opportunity to leverage the ongoing Ohio START initiative and access child welfare-involved families in rural areas, we seek to collect novel, longitudinal activity space and social networks data from 400 families engaging in Ohio START. The study has three specific aims: (1) to determine whether the overlap between parental activity spaces and child welfare workers' referral networks (i.e., proximity and availability of SUD treatment providers) predicts intermediate (i.e., SUD treatment service use, family resilience) and long-term (i.e., parent substance use, child psychosocial-behavioral health, child maltreatment) family health outcomes; (2) to examine how parents' engagement with family peer mentors is associated with changes in the attributes of parental activity spaces and social networks over time and how these changes, in turn, are associated with family health outcomes; (3) to test whether rurality moderates the effects of SUD treatment referral networks, activity spaces, and social networks on family health outcomes. The proposed project will produce valuable knowledge that can be used to modify START and other family-level intervention efforts to mitigate risks and maximize protection in parents' activity spaces and social networks to enhance family resilience, prevent child maltreatment, and promote child well-being in rural communities.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older;
* currently enrolled in Ohio START;
* are unemployed or have family income at or below the federal poverty level,
* designated as the primary parent in the Ohio START case plan.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will include parents who have been impacted by the child welfare system due to co-occurring parental substance use and child maltreatment. Specifically, participants are parents of children of any age between birth and 17 years and 11 months (i.e., less than age 18 years of age) and who have participated in the Ohio Sobriety, Treatment, and Reducing Trauma (Ohio START) intervention. The participant will be 18 years 00 months at minimum. We do not limit the higher end of the participant age. The target sample size for the proposed study is N = 400 parents. In the rare instances where multiple primary parents from the same family are documented, we will randomly select one focal parent (e.g., the parent whose birthday is closest to the referral date).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Parental substance use severity | Baseline, 6 months, and 12 months
  Parental substance use problems will be measured using the Simple Screening Instrument for Alcohol and Other Drugs (SSI-AOD), a 16-item screen that assesses respondents' experiences with substances in the past month and measures the severity of alcohol and other drug problems. In addition, weekly urine drug screening data (tests administered randomly each week) collected from all Ohio START participants will be drawn from the Need Portal and used to objectively assess parental substance use.
Child psychosocial and behavioral health | Baseline, 6 months, and 12 months
  Child psychosocial-behavioral functioning, including emotional symptoms, conduct problems, peer relationships, hyperactivity, prosocial behaviors, and total problems will be assessed using the Strengths and Difficulties Questionnaire (SDQ; 25 items), a well-established brief psychological assessment tool for children 2 to 17 years old. For children ages 2 months to 1 year and 11 months, the Ages & Stages Questionnaires: Social-Emotional (ASQ:SE) will be used.
Child maltreatment | Baseline, 6 months, and 12 months
  Using SACWIS data, we will assess the number of reports made to child protective services (CPS) and the type of maltreatment (e.g., physical, sexual, emotional abuse, neglect).

SECONDARY OUTCOMES:
Substance use disorder (SUD) treatment service use | Baseline, 6-months, and 12-months
  Parents' SUD treatment service utilization (the number of substance use treatment sessions attended) will be measured using the information (e.g., date of the treatment session attended) that behavioral health service providers enter into the Needs Portal.
Family resilience | Baseline, 6 months, and 12 months
  Family resilience score will be computed using the Family Functioning and Resilience subscale of the Protective Factors Survey (PFS; 5 items). Responses on the five items (e.g., "my family pulls together when things are stressful", "my family is able to solve our problems", "in my family, we talk about problems") will be summed to create the total family resilience score.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative Ohio START family survey data generated from the study will be de-identified and shared. The dataset will include three waves of longitudinal data collected at six-month intervals (i.e., Wave 1: baseline, Wave 2: 6-month follow-up, Wave 3: 12-month follow-up) to assess parental activity spaces, social networks, parenting attitudes, family protective factors, and child and family health outcomes. All survey data files will be de-identified before they are archived due to the highly personal and identifiable nature of the target population (i.e., parent enrolled in Ohio START and residing in rural communities) and collected information, such as parental activity spaces (i.e., the name, street, cross-street, city, state, and zip code for each location they frequent for home, school, work, medical care, and child care). Thus, we will de-identify data before sharing data to avoid compromising subject privacy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data and metadata will be made available on Data Sharing for Demographic Research (DSDR) upon their publication or the end of the performance period, whichever comes first. Data and metadata will be available indefinitely.
Access Criteria: Public use data and metadata will be archived in Data Sharing for Demographic Research (DSDR). DSDR is housed within the Inter-university Consortium for Political and Social Research (ICPSR). Data will be findable by the research community in DSDR, which produces a unique DOI for each dataset. We will include our unique DSDR doi number for each publication's data set in publications so that reviewers and readers can locate our data. Publications will be findable by the research community in PubMed through a unique DOI for each publication.

REFERENCES:
- [Background] Young NK, Boles SM, Otero C. Parental substance use disorders and child maltreatment: overlap, gaps, and opportunities. Child Maltreat. 2007 May;12(2):137-49. doi: 10.1177/1077559507300322. PMID 17446567
- [Background] Seay K. How Many Families in Child Welfare Services Are Affected by Parental Substance Use Disorders? A Common Question that Remains Unanswered. Child Welfare. 2015;94(4):19-51. PMID 26827475
- [Background] Norman RE, Byambaa M, De R, Butchart A, Scott J, Vos T. The long-term health consequences of child physical abuse, emotional abuse, and neglect: a systematic review and meta-analysis. PLoS Med. 2012;9(11):e1001349. doi: 10.1371/journal.pmed.1001349. Epub 2012 Nov 27. PMID 23209385
- [Background] Kantor GK, Holt MK, Mebert CJ, Straus MA, Drach KM, Ricci LR, MacAllum CA, Brown W. Development and preliminary psychometric properties of the multidimensional neglectful behavior scale-child report. Child Maltreat. 2004 Nov;9(4):409-28. doi: 10.1177/1077559504269530. PMID 15538039
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Fortney J, Booth BM. Access to substance abuse services in rural areas. Recent Dev Alcohol. 2001;15:177-97. doi: 10.1007/978-0-306-47193-3_10. No abstract available. PMID 11449741